CLINICAL TRIAL: NCT05582902
Title: Longitudinal, App-based Assessment of Varying Red Blood Cell Transfusion Strategies and Their Association With Patient-Reported, Clinical and Economical Outcomes in Lower-risk Myelodysplastic Neoplasms (MDS) Patients
Brief Title: Study Investigating Patient-Reported Outcomes in Lower-risk MDS Patients
Acronym: PRO-RED
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Anne Sophie Kubasch, Principal Investigator, University of Leipzig
Other Study IDs: PRO-RED study
Record Dates: First submitted 2022-09-29; First posted 2022-10-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: MDS; MDS/MPN
Keywords: MDS; anemia; transfusion dependence; quality of life; MDS/MPN
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
PRO-RED is a prospective, longitudinal, and multicenter observational study. Enrolled patients will be followed for 6 months in at least monthly intervals in terms of their received red blood cell transfusions and routine myelodysplastic neoplasms (MDS)-associated clinical parameters. In addition, the participating subjects will be provided with a digital/mobile application covering a smartphone app or paper-based questionnaires to answer a set of quality of life (QoL) questions once a week. During routine visits in the clinical trials center performed by the treating physician (at least every month), patients will answer standardized questionnaires for the assessment of MDS-related QoL. Also, included patients will take a photo of fingernails/eyelids with their smartphone camera with the aim to further analyze these pictures in a way to potentially deduct correlated hemoglobin (Hb)-values. As a long term aim beyond the PRO-RED study, the data will serve as a training cohort for the development of an algorithm for image-based calculation of individual Hb levels.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Confirmed diagnosis of lower-risk myelodysplastic neoplasms (MDS; IPSS-R very low, low, intermediate up to 3.5 points) or MDS/MPN overlap including MDS/MPN-RS-T, MDS/MPNu, aCML or non-proliferative chronic myelomonocytic leukemia (CMML) according to World Health Organization (WHO) criteria as determined by microscopic and standard cytogenetic analyses of the bone marrow and peripheral complete blood count (CBC)
* Symptomatic transfusion dependent (TD) anemia defined as having received ≥3 units of red blood cells (RBC) within the last 16 weeks prior to screening according to the International Working Group (IWG) criteria for MDS (Platzbecker et al. 2019)

Exclusion Criteria:

- Suspected lack of compliance according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from lower-risk myelodysplastic neoplasms (MDS) or MDS/MPN with red blood cell transfusion-dependent anemia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life | 6 months
  health-related quality of life assessed by patient reported questionnaires based on EORTC QLQ-C30
health-related quality of life | 6 months
  health-related quality of life assessed by patient reported questionnaires based on QUALMS
Course of hemoglobin levels | 6 months
  Hemoglobin level measurements at point of care

CONTACTS AND LOCATIONS:
Locations (11):
- Universitätsklinik Innsbruck, Innsbruck, Austria
- Germany (10):
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Jena, Jena
  - University Hospital Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Friedrich-Ebert-Krankenhaus GmbH, Neumünster